CLINICAL TRIAL: NCT00767169
Title: Bisphosphonate-coated Dental Implants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Per Aspenberg, professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tandskruv1
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Edentatio (Toothlessness)
Keywords: Edentatio (Toothlessness)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- coated implant and control (Experimental)
  Interventions: Device: Dental implant coating with a fibrinogen carrier for pamidronate and ibandronate

INTERVENTIONS:
Device: Dental implant coating with a fibrinogen carrier for pamidronate and ibandronate — Dental implant coating with a fibrinogen carrier for pamidronate and ibandronate compared with uncoated controls in the same mouth.

SUMMARY:
Dental implants (screws for fastening false teeth) have been coated with bisphosphonates (drugs that slow down removal of bone). Patients get one such screw and one without coating, by a surgeon who does not know which is which. The screws are compared by measuring how well fixed they are by a vibration measuring technique, and x-rays. The hypothesis is that the bisphosphonates will improve fixation.

ELIGIBILITY:
Inclusion Criteria:

* Need for at least 2 dental implants, which are to be inserted in bone of reasonably similar quality.

Exclusion Criteria:

* Systemic or immunologic disease, alcoholism, uncontrolled diabetes and smoking.
* Local exclusion criteria were: previous tumour, trauma and surgery.
* Also patients with Cawood & Howell class IV - VI maxilla-bone were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Increase in resonance vibration frequency (ISQ units) from insertion to abutment connection as compared to the control in the same patient. | 6 months

SECONDARY OUTCOMES:
Marginal resorption on x-rays | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Per Aspenberg, MD, PhD, Study Chair — Linkoeping University
Locations (1):
- Department of Oral & maxillofacial surgery, University Hospital., Linköping, Sweden

REFERENCES:
- [Result] Abtahi J, Tengvall P, Aspenberg P. A bisphosphonate-coating improves the fixation of metal implants in human bone. A randomized trial of dental implants. Bone. 2012 May;50(5):1148-51. doi: 10.1016/j.bone.2012.02.001. Epub 2012 Feb 10. PMID 22348981